CLINICAL TRIAL: NCT04282629
Title: Efficacy of 10 Days Intravenous Milrinone Treatment to Optimize Cerebral Hemodynamic and Prevent Delayed Cerebral Ischemia (DCI) in Patients with Severe Subarachnoid Hemorrhage Due to Intracranial Aneurysm Rupture
Brief Title: Cerebral Hemodynamic Optimization by Milrinone to Prevent Delayed Cerebral Ischemia
Acronym: OPTIMIL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RC31/18/0472
Record Dates: First submitted 2020-02-17; First posted 2020-02-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Aneurysmal Subarachnoid Hemorrhage
Keywords: Milrinone; Vasospasm; Delayed Cerebral Ischemia
MeSH Terms: conditions — Subarachnoid Hemorrhage | interventions — Milrinone

STUDY DESIGN:
Intervention Model Description: Group milrinone versus group placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Milrinone (Experimental): "milrinone" group benefiting from an identical treatment to the standard care group and in addition, administration of milrinone (0.75 μg / kg / min, intravenous) from Day 4 to Day 14. In case of suspicion of vasospasm and after ineffective effect of medical measures (euvolemia and increase in mean arterial pressure), an endovascular treatment will be possible. The occurrence of vasospasm will be monitored closely with clinical examination and cerebral tissue oxygen pressure (PtiO2). From D4 to D14, general and biological data, clinical examination will be collected daily. Intensive care unit complications (neurologic, pulmonary, cardiac and septic complications) will be collected. At 1 month, the volume of DCI lesions will be measured on CT scan. Neurologic prognosis, quality of life and mortality will be studied at 1 month, 3 month, 6 month and 1 year. Adverse events will be monitored closely.
  Interventions: Drug: Milrinone Injection
- Standard Care (Placebo Comparator): The standard care group will follow the recommended management of SAHa and will receive a placebo (intravenous glucose 5%) from Day 4 to Day 14. In case of suspicion of vasospasm and after ineffective effect of medical measures (euvolemia and increase in mean arterial pressure), an endovascular treatment will be possible. The occurrence of vasospasm will be monitored closely with clinical examination and cerebral tissue oxygen pressure (PtiO2). From D4 to D14, general and biological data, clinical examination will be collected daily. Intensive care unit complications (neurologic, pulmonary, cardiac and septic complications) will be collected. At 1 month, the volume of DCI lesions will be measured on CT scan. Neurologic prognosis, quality of life and mortality will be studied at 1 month, 3 month, 6 month and 1 year. Adverse events will be monitored closely.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Milrinone Injection — administration of milrinone (0.75 μg / kg / min, intravenous) from Day 4 to Day 14
  Arms: Milrinone
Other: Placebo — administration of placebo (intravenous glucose 5%) from Day 4 to Day 14
  Arms: Standard Care

SUMMARY:
The present study is a randomized, multi-center, double-blind, prospective study that tests the efficacy of intravenous milrinone to optimize cerebral hemodynamic and prevent delayed cerebral ischemia (DCI) during the high-risk period (day 4- day 14) in patients with severe subarachnoid hemorrhage due to intracranial aneurysm rupture (SAHa) (WFNS IV-V). The main objective is to evaluate, in comatose patients and / or sedated on D3 following a severe SAHa (WFNS IV -V), the effect of 10 days of milrinone versus placebo, in addition to the usual management, on the volume of DCI lesions measured on CT scan at 1 month.

DETAILED DESCRIPTION:
After SAHa, approximately 28% of patients will present DCI. DCI is a major cause of death and disability and will condition the neurological prognosis. Its treatment is not really codified, because of the absence of scientific proof of good level. Milrinone, an inhibitor of type III phosphodiesterase, seems particularly interesting in the management of DCI. This molecule has indeed a powerful vasodilator action. In addition, its anti-inflammatory effects could inhibit the abnormal proliferation of vascular smooth muscle cells and the remodelling observed in patients with DCI via an action on interleukin-6. Finally, because of its positive inotropic effect, it is an interesting choice in these patients with neurogenic cardiomyopathy where the administration of catecholamines is to be avoided. Strong evidence for efficacy of milrinone in the treatment and / or prevention of DCI is still lacking. All patients will benefit from a computed tomography (CT) brain imaging at 48 hrs following aneurysm treatment to define baseline imaging. The standard care (SC) group will follow the recommended management of SAHa and will receive a placebo (intravenous glucose 5%) from day 4 to day 14. The milrinone (M) group will receive, in addition to standard care, administration of milrinone (0.75 μg / kg / min, intravenous) from day 4 to day 14. In case of suspicion of vasospasm and after ineffective effect of medical measures (euvolemia and increase in mean arterial pressure), an endovascular treatment will be possible. The occurrence of vasospasm will be monitored closely with clinical examination and cerebral tissue oxygen pressure (PtiO2). From day 4 to day 14, general and biological data, clinical examination will be collected daily. Intensive care unit complications (neurologic, pulmonary, cardiac and septic complications) will be collected. At 1 month, the volume of DCI lesions will be measured on CT scan. Neurologic prognosis, quality of life and mortality will be studied at 1 month, 3 month, 6 month and 1 year. Adverse events will be monitored closely.

ELIGIBILITY:
Inclusion Criteria:

* patients with severe SAHa (WFNS IV and V,) whose neurological examination is impossible because of coma (Glasgow coma score of 8 or less) or need for sedation at D3
* absence of pre-existing neurological handicap (mRS 0-2)
* major patient (≥ 18 years)
* affiliation to social security or benefiting through a third person
* free patient, without tutorship or curatorship or under judicial protection
* obtaining a signed informed consent by a relative (or the person of trust) after clear and fair information about the study.

Exclusion Criteria:

* patients with non-severe SAHa (WFNS I, II and III)
* Occurrence of a major complication (haemorrhagic or ischaemic) documented during the procedure of securing the aneurysm and endangering the short-term vital prognosis
* heart failure requiring inotropic administration at the time of randomization
* ICHT at the time of randomisation (ICP> 25 mmHg for at least 20 min)
* known severe obstructive heart diseases
* flutter patient or atrial fibrillation
* hypotension and / or severe hypovolemia with hemodynamic instability
* septic shock
* acute / chronic renal insufficiency (Cl <50ml / min)
* major hydroelectrolytic disorders (hypokalemia <3 mmol / L)
* known hypersensitivity to milrinone or any of the excipients
* early limitation of life-sustaining care
* pregnancy, breastfeeding
* permanent contraindications to MRI
* participation in another clinical interventional study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Estimated)
Dates: Start 2021-07-25 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
volume of delayed cerebral ischemia lesions | 1 month
  volume of DCI lesions measured on CT scan and validated by Magnetic Resonance Imaging (MRI) imaging at 1 month

SECONDARY OUTCOMES:
Radiological parameters on CT at 1 month | 1 month
  percentage of patients with DCI lesions
Evolution in intensive care: Neurological complications 1 | 1 month
  number of episodes of PtiO2 below the ischemic threshold in intensive care: PtiO2 <20 mmHg (moderate hypoxia) and <15 mm Hg (severe hypoxia) for at least 15 minutes
Evolution in intensive care: Neurological complications 2 | 1 month
  total duration of episodes of PtiO2 <20 mm Hg (moderate hypoxia) and <15 mm Hg (severe hypoxia)
Evolution in intensive care: Neurological complications 3 | 1 month
  number of recourse to an endovascular treatment
Evolution in intensive care: Neurological complications 4 | 1 month
  intracranial hypertension in intensive care: ICP> 20 mmHg for at least 15 minutes.
Number and type of non-neurological complications | 1 month
  non-neurological complications
Number of days in intensive care | 1 month
  Number of days in intensive care
Number of days with mechanical ventilation | 1 month
  Number of days with mechanical ventilation
neurological prognosis at 1 month: Rankin score | 1 month
  evaluated by the modified Rankin score (good prognosis: mRS 0, 1 and 2 / poor prognosis: mRS 3, 4 and 5)
neurological prognosis at 1 month: Glasgow Outcome scale | 1 month
  evaluated by the Glasgow Outcome Scale (GOS) (good prognosis: GOS 4 and 5 / poor prognosis: GOS 1, 2 and 3).
neurological prognosis at 3 month: Rankin score | 3 month
  evaluated by the modified Rankin score (good prognosis: mRS 0, 1 and 2 / poor prognosis: mRS 3, 4 and 5)
neurological prognosis at 3 month: Glasgow Outcome scale | 3 month
  evaluated by the the Glasgow Outcome Scale (good prognosis: GOS 4 and 5 / poor prognosis: GOS 1, 2 and 3)
neurological prognosis at 6 month: Rankin score | 6 month
  evaluated by the modified Rankin score (good prognosis: mRS 0, 1 and 2 / poor prognosis: mRS 3, 4 and 5)
neurological prognosis at 6 month: Glasgow Outcome scale | 6 month
  evaluated by the the Glasgow Outcome Scale (good prognosis: GOS 4 and 5 / poor prognosis: GOS 1, 2 and 3)
neurological prognosis at 1 year: Rankin score | 1 year
  evaluated by the modified Rankin score (good prognosis: mRS 0, 1 and 2 / poor prognosis: mRS 3, 4 and 5)
neurological prognosis at 1 year: Glasgow Outcome scale | 1 year
  evaluated by the Glasgow Outcome Scale (good prognosis: GOS 4 and 5 / poor prognosis: GOS 1, 2 and 3)
Mortality at 1 month | 1 month
  Mortality at 1 month
Mortality at 3 month | 3 month
  Mortality at 3 month
Mortality at 6 month | 6 month
  Mortality at 6 month
Mortality at 1 year | 1 year
  Mortality at 1 year
number of days of hospitalization | 1 year
  number of days of hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Geeraerts, MD PhD, Principal Investigator — University Hospital, Toulouse
Locations (5):
- France (5):
  - University Hospital Bordeaux, Bordeaux
  - CHUGA, Grenoble
  - University Hospital of La Réunion, La Réunion
  - HCL, Lyon
  - University Hospital of Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No